CLINICAL TRIAL: NCT05364918
Title: Clinical Effect Of Application Of Jeksung Combined With Anti-radiation Spray In Patients Radiotherapy-Induced Oral Mucositis Of Local Advanced Head And Neck Tumors
Brief Title: Clinical Study On Acute Radiotherapy-Induced Oral Mucositis In Patients With Locally Advanced Head And Neck Tumors
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Radioactive Oral Mucositis
Record Dates: First submitted 2022-04-28; First posted 2022-05-06 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2020-08

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Jeksung (Experimental)
  Interventions: Drug: Jeksung combined with anti-radiation spray
- Control (No Intervention)

INTERVENTIONS:
Drug: Jeksung combined with anti-radiation spray — Treat radiation stomatitis with Jeksung combined with anti-radiation spray
  Arms: Jeksung

SUMMARY:
To explore a more efficient and scientific clinical treatment plan for acute radiotherapy-induced oral mucositis(RIOM/RTOM).it is hoped that the drug combination can more effectively improve the cure rate of acute RIOM,reduce the degree of oral mucosal injury and utilization rate of analgesic drugs,and reduce the occurrence of severe acute RIOM. Almost all patients with head and neck will have RIOM because of receiving radiation therapy.Studies have shown that the incidence of severe acute RIOM accounted for about 34% to 56%.There is no specific drug when acute RIOM is often accompanied by varying degrees of pain and infection in the mouth.Severe RIOM seriously affects ingestion through the mouth and doesn't conducive to the treatment and prognosis of tumor diseases. To further explore the efficiency and advantages of the combined application of Jeksung and anti-radiation spray in the treatment of acute RIOM at all levels,and provide more data support for relevant clinical treatment.Explore whether the Jeksung with combination of anti-radiation spray can effectively delay the occurrence of acute RIOM and delay the course of the disease.It will be expected to improve the quality of life of cancer patients ,reduce the occurrence of adverse events due during radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Head and neck cancer was confirmed by patholog
* Received radical radiotherapy, and were observed and treated by RTOM in the stomatology department
* Age range: 18-75 years old
* The estimated survival period is more than 6 months, and the card functional status score (KPS) is 70
* There are no diseases that affect the treatment of oral mucositis, such as mouth opening restriction, Sjogren's syndrome, etc.
* Sign the informed consent form

Exclusion Criteria:

* Failed to complete radiotherapy, or delayed radiotherapy more than 2 weeks than planned
* There are previous oral mucosal diseases, such as oral lichen planus and pemphigus, which are not effectively controlled or still need long-term drug treatment
* There are other diseases that affect radiotherapy, such as severe organ function injury, chronic infectious diseases, etc.
* Had received radiotherapy for head and neck for other diseases;
* The expected survival time is less than 6 months;
* Refuse to provide personal information or sign informed consent
* The investigator judged other conditions that might affect the conduct of the clinical study and the determination of the study results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-08-17 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Acute radiotherapy-induced oral mucositis | The first day of radiation therapy for head and neck tumors to the last day
  Occur rate of severe radiotherapy-induced oral mucositis

SECONDARY OUTCOMES:
Oral pain | The first day to the last day of radiation therapy for head and neck tumors
  Utilization rate of analgesic drugs

CONTACTS AND LOCATIONS:
Overall Officials: Yu Zeng, Dr., Principal Investigator — Affiliated Cancer Hospital & Institute of Guangzhou Medical University
Locations (1):
- Yu Zeng, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No